CLINICAL TRIAL: NCT02995603
Title: Nano-X: Patient Experience and Acceptance of Horizontal Rotation
Brief Title: Patient Experience and Acceptance of Horizontal Rotation
Acronym: Nano-X
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Prince of Wales Hospital, Sydney (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Nano-X V1
Record Dates: First submitted 2016-12-07; First posted 2016-12-16 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cancer
Keywords: Radiotherapy; Rotation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient rotation (Experimental): Patients will be rotated horizontally, using the Nano-X patient rotation system, and asked to complete validated questionnaires to quantify their experience.
  Interventions: Device: Nano-X patient rotation

INTERVENTIONS:
Device: Nano-X patient rotation — Patients are required to completed validated questionnaires to quantify their experience of horizontal rotation.

SUMMARY:
Patients will complete validated psychometric questionnaires to quantify their experience of being rotated at different speeds using the Nano-X patient rotation system.

DETAILED DESCRIPTION:
Study participants will be asked to attend the clinic on two separate occasions. Each session will last less than one hour. Patients will be asked to complete validated psychometric surveys assessing 1) their level of claustrophobia, 2) their level of anxiety and 3) their (baseline) motion sickness, before and after each session. They will then be rotated 3-4 times on the Nano-X patient rotation system, at varying speeds ranging from 6°/sec to 45°/sec. Each rotation will be designed to simulate a typical radiotherapy treatment; that is 9 angles, pausing for around 30 seconds at each angle. Straight after each rotation, patients will again complete the questionnaire assessing their anxiety levels and motion sickness.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of cancer, any stage
2. ≥18 years of age
3. Eastern Cooperative Oncology Group (ECOG) status 0-2
4. Currently or previously being treated with radiotherapy
5. Any prior therapy allowed
6. Willing and able to comply with all study requirements
7. Must be able to read and complete questionnaires in English
8. Signed, written informed consent

Exclusion Criteria:

1. Pregnant women
2. Mentally impaired patients or patients for whom attaining informed consent would be difficult (including language barriers)
3. Severe vertigo or recent diagnosis of Benign Paroxysmal Positioning Vertigo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in level of patient anxiety following rotation in the Nano-X Patient Rotation System | 1 hour
  Comparison of mean scores of Short Form State/Trait Anxiety Inventory (STAI) Questionnaire outcomes before and after being rotated in the Nano-X Patient Rotation System
Change in level of patient motion sickness following rotation in the Nano-X Patient Rotation System | 1 hour
  Comparison of mean scores of Fast Motion Sickness Test (FMS) Questionnaire outcomes before and after being rotated in the Nano-X Patient Rotation
Correlation between claustrophobia and the change in anxiety and motion sickness of patients following rotation in the Nano-X Patient Rotation System | 1 year
  Correlation between Claustrophobia Questionnaire (CLQ) scores prior to study participation on the anxiety and motion sickness results measured in Outcome 1 and Outcome 2

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keall, Prof, Study Chair — University of Sydney
Locations (1):
- Prince of Wales Hospital, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No